CLINICAL TRIAL: NCT07101978
Title: Influence of Serial Whole-body Hyperthermia on Circadian Core Body Temperature, the Somatosensory System and Movement Evoked Pain: Differences Between Healthy Subjects and Patients With Chronic Primary Pain
Brief Title: Hyperthermia in Patients With Chronic Primary Pain - Effects on Thermoregulation, Somatosensory System and Movement Evoked Pain
Acronym: HYPPRI-1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bern University of Applied Sciences (Other)
Collaborators: Dr. med. h.c Erwin Braun Stiftung (Unknown)
Responsible Party: Principal Investigator, Kay-Uwe Hanusch, Principal Investigator,, Bern University of Applied Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F.016677-42-PHYW-1
Record Dates: First submitted 2025-07-08; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Hyperthermia; Chronic Primary Pain; Widespread Pain; Muscular Disease; Rheumatic Diseases; Musculoskeletal Diseases; Neuromuscular Disease; Fibromyalgia; Circadian Rhythm; Body Temperature Changes; Somatosensory Function; Quantitative Sensory Testing; Healthy
Keywords: hyperthermia; widespread pain; chronic primary pain; circadian body temperature; quantitative sensory testing; healthy
MeSH Terms: conditions — Hyperthermia; Chronic Pain; Muscular Diseases; Rheumatic Diseases; Musculoskeletal Diseases; Neuromuscular Diseases; Fibromyalgia; Body Temperature Changes

STUDY DESIGN:
Intervention Model Description: Quasi-experimental pre-post study design with a healthy and a patients group with the the same intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- serial whole body hyperthermia (Experimental): For the study, the method of water-filtered whole-body hyperthermia is used. The HT 3000 system (by heckel medizintechnik GmbH, Olgastrasse 25, 73728 Esslingen, Garmany) is used, in which the entire body is heated to a core body temperature above the physiological 37°C. The aim is to achieve a core body temperature of 38.5°C within the framework of mild whole-body hyperthermia. After this warm-up phase, a temperature plateau phase of about 15 minutes follows, in which an attempt is made to maintain the core body temperature of 38.5°C. In the temperature plateau phase, a slight increase in the body core temperature is usually observed. The total time required for a session is given as 2.5 to 3 hours, but this depends on the individual constitution and daily condition of the patient and can be subject to fluctuations.
  Interventions: Behavioral: serial whole body hyperthermia

INTERVENTIONS:
Behavioral: serial whole body hyperthermia — The hyperthermia treatment is carried out in a cycle of two treatments per week, with at least one day in between, over a period of three weeks, according to the manufacturer's instructions. According to the guidelines, the rectal (possibly vaginal) temperature (as body core temperature), heart rate and oxygen saturation (Sp02) are continuously determined during the hyperthermiatreatment. During the treatment, continuous supervision by trained personnel is guaranteed, and a doctor is on call.
  Other Names: passive whole body hyperthermia; water filtered whole body hyperthermia; moderate whole body infrared-A hyperthermia

SUMMARY:
This study, in a quasi-experimental pre-post design, investigates the effect of serial water-filtered whole-body hyperthermia on circadian core body temperature, the somatosensory system (nociception) and pain perception in healthy and patients with chronic primary pain (e.g., fibromyalgia). The intervention lasts 3 weeks with two treatment sessions per week.

DETAILED DESCRIPTION:
A total of 30 healthy participants and 30 participants with chronic primary pain between the ages of 18 and 70 are being sought. All participants will receive the same amount of water-filtered whole-body hyperthermia in outpatient or semi-inpatient treatment. All abnormalities and side effects will be documented by the responsible therapists and doctors. Changes in circadian core body temperature, sensory or nociceptive sensitivities of the somatosensory system, and movement-evoked pain will be recorded, and blood parameters for nociceptive plasticity will be collected. For secondary efficacy, specific questionnaires on pain experience, fatigue, depression, and fear avoidance behavior will be collected 7 and 25 weeks after therapy.

ELIGIBILITY:
Inclusion Criteria:

patients:

* Confirmed diagnosis of widespread pain (ICD-11 MG30.01)
* Widespread Pain Index (WPI) ≥ 7 and Symptom Severity (SS) scale ≥ 5 or WPI) ≥ 3 and SS ≥ 9,
* Pain >= 3 month and VAS >= 4,0
* Body - infrared-A-Bulb Distance < 38cm (overweight participants)
* Signed declaration of consent

healthy:

* No chronic illnesses
* No acute infections
* No regular medication: To avoid interactions
* BMI ≤ 40kg/cm2
* Mental health: No psychiatric diagnoses or psychotropic medication in your medical history

Exclusion Criteria:

* Participation in other clinical studies
* Contraindications for hyperthermia (severe cardiovascular diseases, tumour diseases, acute infections, pregnant and breastfeeding women)
* Acute and / or feverish microbial infections
* Participants with severe somatic, rheumatic concomitant endocrine or neurological diseases, in particular neurological diseases associated with cognitive disorders, severe liver or kidney and cardiac diseases
* participants who are permanently treated with opioids, cannabis, immunosuppressive drugs (e.g. corticoids, immunosuppressants) or alpha/beta-A(nta)gonists due to a disease from the group described above
* participants with pain due to a serious psychiatric illness (bipolar disorder, psychosis, personality disorder, severe depression, substance abuse) and serious systemic or neurological disorders
* pregnancy or breastfeeding (for women)
* Intake of medication within 6 weeks that inhibits the reuptake of the neurotransmitter serotonin or binds to receptors of this neurotransmitter group

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Circadian core body temperature | Week 0
  A BodyCap HF (high-frequency) measurement capsule is used for circadian monitoring of core body temperature over a 24-hour period. The single-use capsule is swallowed and excreted naturally after the measurement.
Circadian core body temperature | Week 5
  A BodyCap HF (high-frequency) measurement capsule is used for circadian monitoring of core body temperature over a 24-hour period. The single-use capsule is swallowed and excreted naturally after the measurement.
Cold detection threshold (CDT); °C | Week 0
  CDT is a part of quantitative sensory testing. A psychophysical testing method in which calibrated cold temperature stimuli (Thermode) 3x applied to the skin. Z-values are calculate.
Cold detection threshold (CDT); °C | week 5
  CDT is a part of quantitative sensory testing. A psychophysical testing method in which calibrated cold temperature stimuli (Thermode) 3x applied to the skin. Z-values are calculate.
Warm detection threshold (WDT); °C | Week 0
  WDT is a part of quantitative sensory testing. A psychophysical testing method in which calibrated warm temperature stimuli (Thermode) 3x applied to the skin. Z-values are calculate.
Warm detection threshold (WDT); °C | week 5
  WDT is a part of quantitative sensory testing. A psychophysical testing method in which calibrated warm temperature stimuli (Thermode) 3x applied to the skin. Z-values are calculate.
Thermal sensory limen (TSL) ; °C | week 0
  TSL is a part of quantitative sensory testing. A psychophysical testing method in which calibrated warm and cold temperature stimuli (Thermode) alternately 6x applied to the skin. Z-values are calculate and count number of cold stimuli that are perceived as hot.
Thermal sensory limen (TSL) ; °C | week 5
  TSL is a part of quantitative sensory testing. A psychophysical testing method in which calibrated warm and cold temperature stimuli (Thermode) alternately 6x applied to the skin. Z-values are calculate and count number of cold stimuli that are perceived as hot.
Cold pain threshold (CPT); °C | week 0
  CPT is a part of quantitative sensory testing. A psychophysical testing method in which calibrated nociceptive cold temperature stimuli (Thermode) 3x applied to the skin. Z-values are calculate.
Cold pain threshold (CPT); °C | week 5
  CPT is a part of quantitative sensory testing. A psychophysical testing method in which calibrated nociceptive cold temperature stimuli (Thermode) 3x applied to the skin. Z-values are calculate.
Heat pain threshold (HPT); °C | week 0
  HPT is a part of quantitative sensory testing. A psychophysical testing method in which calibrated nociceptive heat temperature stimuli (Thermode) 3x applied to the skin. Z-values are calculate.
Heat pain threshold (HPT); °C | week 5
  HPT is a part of quantitative sensory testing. A psychophysical testing method in which calibrated nociceptive heat temperature stimuli (Thermode) 3x applied to the skin. Z-values are calculate.
Mechanical detection threshold (MDT) ; mN | week 0
  MDT is a part of quantitative sensory testing. A psychophysical testing method in which calibrated mechanical stimuli (different strengths Frey filaments) 10x applied to the skin Z-values are calculated.
Mechanical detection threshold (MDT) ; mN | week 5
  MDT is a part of quantitative sensory testing. A psychophysical testing method in which calibrated mechanical stimuli (different strengths Frey filaments) 10x applied to the skin Z-values are calculated.
Mechanical pain threshold (MPT), count of sharp and blunt stimuli | week 0
  MPT is a part of quantitative sensory testing. A psychophysical testing method in which calibrated mechanical stimuli (PinPrick with different weights) 10x applied to the skin. Mechanical pain threshold (MPT). Count number of sharp and blunt stimuli. Z-values are calculated.
Mechanical pain threshold (MPT), count of sharp and blunt stimuli | week 5
  MPT is a part of quantitative sensory testing. A psychophysical testing method in which calibrated mechanical stimuli (PinPrick with different weights) 10x applied to the skin. Mechanical pain threshold (MPT). Count number of sharp and blunt stimuli. Z-values are calculated.
Mechanical pain sensitivity (MPS) ; NRS | week 0
  MPS is a part of quantitative sensory testing. A psychophysical testing method in which calibrated mechanical stimuli (PinPrick with different weights) 35x applied to the skin. The Numeric Rating Scale (0 = no pain to 100 = worst pain imaginable) is queried. Z-values are calculated.
Mechanical pain sensitivity (MPS) ; NRS | week 5
  MPS is a part of quantitative sensory testing. A psychophysical testing method in which calibrated mechanical stimuli (PinPrick with different weights) 35x applied to the skin. The Numeric Rating Scale (0 = no pain to 100 = worst pain imaginable) is queried. Z-values are calculated.
Summative pain amplification (WUR); NRS | week 0
  WUR (wind-up ratio) is a part of quantitative sensory testing. A psychophysical testing method in which calibrated mechanical stimuli (PinPrick with different weights) single and seriell 10x applied to the skin. The Numeric Rating Scale (0 = no pain to 100 = worst pain imaginable) for single and seriell stimuli are compared into relation. Z-values are calculated.
Summative pain amplification (WUR); NRS | week 5
  WUR (wind-up ratio) is a part of quantitative sensory testing. A psychophysical testing method in which calibrated mechanical stimuli (PinPrick with different weights) single and seriell 10x applied to the skin. The Numeric Rating Scale (0 = no pain to 100 = worst pain imaginable) for single and seriell stimuli are compared into relation. Z-values are calculated.
Vibration detection threshold (VDT) ; x/8 | week 0
  VDT is a part of quantitative sensory testing. A psychophysical testing method in which calibrated mechanical stimuli (64Hz tuning fork) 3x applied to the skin. The x/8 vibration is measure (0/8 no perception and 8/8 strengthest perception). Z-values are calculated.
Vibration detection threshold (VDT) ; x/8 | week 5
  VDT is a part of quantitative sensory testing. A psychophysical testing method in which calibrated mechanical stimuli (64Hz tuning fork) 3x applied to the skin. The x/8 vibration is measure (0/8 no perception and 8/8 strengthest perception). Z-values are calculated.
Pressure pain threshold (PPT), kgf/1cm2 | week 0
  PPT is a part of quantitative sensory testing. A psychophysical testing method in which calibrated mechanical stimuli (pain pressure algometer) 5x applied to the skin. Z-values are calculated.
Pressure pain threshold (PPT), kgf/1cm2 | week 5
  PPT is a part of quantitative sensory testing. A psychophysical testing method in which calibrated mechanical stimuli (pain pressure algometer) 5x applied to the skin. Z-values are calculated.
Dynamic mechanical allodynia (DMA), NRS | week 0
  DMA is a part of quantitative sensory testing. A psychophysical testing method in which calibrated mechanical stimuli (brush, cotton wool and Q-Tip) 5x applied to the skin. Z-values are calculated. The Numeric Rating Scale (0 = no pain to 100 = worst pain imaginable) ist queried. Z-values are calculated.
Dynamic mechanical allodynia (DMA), NRS | week 5
  DMA is a part of quantitative sensory testing. A psychophysical testing method in which calibrated mechanical stimuli (brush, cotton wool and Q-Tip) 5x applied to the skin. Z-values are calculated. The Numeric Rating Scale (0 = no pain to 100 = worst pain imaginable) ist queried. Z-values are calculated.
6-Minute Walk Test (6MWT) | Week 0
  Walking back and forth as far as possible along a 30-meter corridor in 6 minutes, taking breaks as needed ( total distance covered is recorded in meters, pain is measured before and after the test, 0 = no pain, 10 = worst pain imaginable)
6-Minute Walk Test (6MWT) | Week 5
  Walking back and forth as far as possible along a 30-meter corridor in 6 minutes, taking breaks as needed ( total distance covered is recorded in meters, pain is measured before and after the test, 0 = no pain, 10 = worst pain imaginable)

SECONDARY OUTCOMES:
McGill Pain Questionnaire (MPQ) | Week 0
  The instrument assesses subjective pain experience and evaluates both the quality and numerical intensity of pain (0 = no pain; 10 = worst pain imaginable)
McGill Pain Questionnaire (MPQ) | Week 5
  The instrument assesses subjective pain experience and evaluates both the quality and numerical intensity of pain (0 = no pain; 10 = worst pain imaginable)
McGill Pain Questionnaire (MPQ) | Week 12
  The instrument assesses subjective pain experience and evaluates both the quality and numerical intensity of pain (0 = no pain; 10 = worst pain imaginable)
McGill Pain Questionnaire (MPQ) | Week 30
  The instrument assesses subjective pain experience and evaluates both the quality and numerical intensity of pain (0 = no pain; 10 = worst pain imaginable)
TAMPA-Scale (Kinesiophobia) | Week 0
  Is a psychological questionnaire designed to measure a person's fear of movement and (re)injury due to physical activity. 17 items on a 4-point Likert scale (from "strongly disagree" to "strongly agree
TAMPA-Scale (Kinesiophobia) | Week 5
  Is a psychological questionnaire designed to measure a person's fear of movement and (re)injury due to physical activity. 17 items on a 4-point Likert scale (from "strongly disagree" to "strongly agree
TAMPA-Scale (Kinesiophobia) | Week 12
  Is a psychological questionnaire designed to measure a person's fear of movement and (re)injury due to physical activity. 17 items on a 4-point Likert scale (from "strongly disagree" to "strongly agree
TAMPA-Scale (Kinesiophobia) | Week 30
  Is a psychological questionnaire designed to measure a person's fear of movement and (re)injury due to physical activity. 17 items on a 4-point Likert scale (from "strongly disagree" to "strongly agree
Multidimensional Fatigue Inventory (MFI-20) | Week 0
  An inventory including 20 questions about fatigue-symptoms (each from 1 ("Yes, that is true") to 5 ("No, that is not true")) covering 5 dimensions (general fatigue, physical fatigue, reduced motivation, reduced activity, mental fatigue)
Multidimensional Fatigue Inventory (MFI-20) | Week 5
  An inventory including 20 questions about fatigue-symptoms (each from 1 ("Yes, that is true") to 5 ("No, that is not true")) covering 5 dimensions (general fatigue, physical fatigue, reduced motivation, reduced activity, mental fatigue)
Multidimensional Fatigue Inventory (MFI-20) | Week 12
  An inventory including 20 questions about fatigue-symptoms (each from 1 ("Yes, that is true") to 5 ("No, that is not true")) covering 5 dimensions (general fatigue, physical fatigue, reduced motivation, reduced activity, mental fatigue)
Multidimensional Fatigue Inventory (MFI-20) | Week 30
  An inventory including 20 questions about fatigue-symptoms (each from 1 ("Yes, that is true") to 5 ("No, that is not true")) covering 5 dimensions (general fatigue, physical fatigue, reduced motivation, reduced activity, mental fatigue)
General Depression Scale (ADS-L) | Week 0
  is a german self-report questionnaire designed to assess depressive symptoms in the general population adapted from the CES-D. (20 items, 4-point Likert scale (0 = rarely or none of the time, 3 = most or all of the time)
General Depression Scale (ADS-L) | Week 5
  is a german self-report questionnaire designed to assess depressive symptoms in the general population adapted from the CES-D. (20 items, 4-point Likert scale (0 = rarely or none of the time, 3 = most or all of the time)
General Depression Scale (ADS-L) | Week 12
  is a german self-report questionnaire designed to assess depressive symptoms in the general population adapted from the CES-D. (20 items, 4-point Likert scale (0 = rarely or none of the time, 3 = most or all of the time)
General Depression Scale (ADS-L) | Week 30
  is a german self-report questionnaire designed to assess depressive symptoms in the general population adapted from the CES-D. (20 items, 4-point Likert scale (0 = rarely or none of the time, 3 = most or all of the time)

OTHER OUTCOMES:
BDNF | Week 0
  Brain-Derived Neurotrophic Factor (BDNF) in blood to measure nociplasticity
BDNF | Week 5
  Brain-Derived Neurotrophic Factor (BDNF) in blood to measure nociplasticity
PRISE (Patient-Rated Inventory of Side Effects) | 30min post treatment
  A tool used to assess the presence and severity of side effects (0=no severity, 3= greater severity) across nine organ/function domains, including gastrointestinal, nervous system, heart, eyes/ears, skin, genital/urinary, sleep, sexual function, and other areas

CONTACTS AND LOCATIONS:
Overall Officials: Kay-Uwe Hanusch, Dr.scient.med, Study Director — Bern University of Applied Sciences
Locations (1):
- Bern University of Applied Science, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No